CLINICAL TRIAL: NCT02667470
Title: Overactive Bladder Symptom Scores (OABSS) Responsiveness Before and After Anticholinergic Treatment in Women With Overactive Bladder (OAB)
Brief Title: Reproducibility Study of OABSS and Its Response to Treatment
Acronym: RESORT part 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATH-002
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Overactive Bladder
Keywords: Solifenacin; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solifenacin (Experimental)
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — Oral
  Other Names: Vesicare

SUMMARY:
The objective of this study is to evaluate change of Overactive Bladder (OAB) Symptom Score (OABSS) scores between before and after Solifenacin treatment to OAB patients and to evaluate correlation between change of OABSS scores and other measures for OAB symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At screening visit (Week -2):

  * Symptoms of OAB ≥ 3 months
  * Number of urgency episodes in last 3 days ≥ 3
* Based on the 3-day micturition diary prior to Visit 1 (Week 0):

  * Number of micturition per day ≥ 8
  * Number of urgency episodes in 3 days ≥ 3

Exclusion Criteria:

* At screening visit (Week -2):

  * Stress is the predominant factor as determined by the investigator
  * Indwelling catheters or practicing intermittent self-catheterization
  * Symptomatic urinary tract infection, chronic inflammation
  * Treatment for OAB was started, quitted or changed in 4 weeks
  * Diabetic neuropathy
* At Visit 1 (Week 0):

  * Patient who did not complete the 3-day micturition diary according to the instruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in OABSS scores from prior to treatment and after treatment | Prior to treatment and after treatment (up to 12 weeks)

SECONDARY OUTCOMES:
Correlation of change between OABSS scores and number of micturitions per day | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and number of incontinence episodes per day | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and number of urgency episodes per day | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and number of nocturia episodes per day | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and number of total voided volume per day | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and number of pads per day | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and total International Prostate Symptom Score (IPSS) score | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and IPSS Quality of Life (QoL) score | Prior to treatment and after treatment (up to 12 weeks)
Correlation of change between OABSS scores and Patient Perception of Bladder Condition (PPBC) total score | Prior to treatment and after treatment (up to 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site: 1, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided